CLINICAL TRIAL: NCT02217358
Title: Value of Narrow Band Imaging (NBI) Endoscopy in the Early Diagnosis of Laryngeal Cancer and Precancerous Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FNO-ENT-NBI; RVO - FNOs/2012 (Other Grant/Funding Number: Institutional Support, Ministry of Health, Czech Republic)
Record Dates: First submitted 2014-07-31; First posted 2014-08-15 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Inflammation of Hypopharynx; Hoarseness; Macroscopic Laryngeal Lesions; Histological Confirmation of Dysplasia; Carcinoma in Situ; Invasive Carcinoma of Larynx; Invasive Carcinoma of Hypo Pharynx; Recurrent Respiratory Papillomatosis
Keywords: squamous cell carcinoma of the head and neck; NBI endoscopy; videoendoscopy; white light endoscopy; magnifying endoscopy; direct laryngoscopy
MeSH Terms: conditions — Hoarseness; Carcinoma in Situ; Recurrent respiratory papillomatosis; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NBI endoscopy (Experimental): 150 patients with suspected lesion in larynx and hypopharynx on standard ENT white light endoscopy examination will undergo NBI endoscopy in order to compare the outcomes of these two examination methods
  Interventions: Device: NBI endoscopy

INTERVENTIONS:
Device: NBI endoscopy — see in "detail description of the study" part of the protocol

SUMMARY:
The aim of the project is to compare NBI endoscopy and standard endoscopic method using white light and evaluate accuracy both methods in early detection and diagnosis hypopharyngeal and laryngeal precancerous and cancerous lesions. A higher contrast between the mucosal epithelium and blood vessels is achieved in NBI endoscopy using filtered light comparing to white light observations. This allows detection of small mucosal changes, few millimetres in diameter, which are not observable using white light. The second aim in patients with squamous cell carcinoma of the upper aerodigestive tract is to compare extension of mucosal lesions by evaluation of NBI endoscopy and white light endoscopy, which is crucial for perform targeted biopsy and for determination of resection margins in cancer surgery. The investigators expect that dysplastic changes of mucosa or early laryngeal cancerous lesions are detected in white light endoscopy rarely. In case our hypothesis is confirmed, frequency of precancerous and early cancerous lesions of hypopharynx and larynx is more common in patients with non-specific symptoms of laryngeal and pharyngeal diseases.

DETAILED DESCRIPTION:
Laryngeal squamous cell carcinoma (SCC) is one of the most common head and neck cancers. In many cases laryngeal SCC is diagnosed too late for curative treatment - the reasons are non-specific symptoms and very often poor social status of patients, on the other hand also limited diagnostics modalities. Its early detection and diagnosis is essential in order to maximise cure rates and to preserve vocal function. Radiological evaluation with computer tomography (CT) and magnetic resonance imaging (MRI) provides vital information on the extent of the primary tumor and the presence of cervical lymph node metastasis, but fails to identify superficial mucosal abnormalities. At present, white light laryngoscopy combined with biopsy is the standard diagnostic procedure in the assessment of laryngeal cancer and precancerous lesions. However, white light laryngoscopy provides poor quality images and has difficulty identifying epithelial changes and directly differentiating benign from malignant tumors in vivo.

The best case scenario for early detection of SCC of the upper aerodigestive tract (UADT) would be at the stage of squamous dysplasia or even carcinoma in situ. These early lesions are very difficult to detect even with multiple passes with the endoscope, if they are ≤ 1 cm in diameter. In gastroenterology are still more common used endoscopies with high magnification for detection pathological mucosal lesions, but in otorhinolaryngology is using these equipments still limited. However, in recent years are detected epithelial lesions more common by biological endoscopic methods. A well established technique, already in use for the oesophagus, is Lugol chromoendoscopy, where squamous dysplasia and carcinoma in situ appear as Lugol voiding lesions (Watanabe et al., 2003). These precancerous lesions can be easily resected via endoscopic mucosal resection, which is a minimally invasive procedure with short hospital stay. However, this technique cannot be applied in the head and neck region due to the severe mucosal irritation that may lead to severe dysphagia and even aspiration. Other biological endoscopic methods include autofluorescence, contact endoscopy or narrow band imaging.

Recently, a new high-resolution endoscopic technique, narrow band imaging, has begun to be widely used in the early diagnosis of gastrointestinal cancer. Narrow band imaging is based upon the fact that the depth of light penetration depends on the light wavelength: the longer the wavelength, the deeper the penetration. Narrow band imaging modifies the broadband white light from a xenon lamp into two narrow band illumination beams with central wavelengths of 415nm - blue light, which is designed to primarily penetrate the musoca and display superficial capillary networks, and 540 nm - green light designed to penetrate the submucosa and visualized subepithelial vessels. When these two wavelengths are used in combination, they provide and extremely high contrast image of the tissue surface. In literature (Ni et al., 2011) is described classification of intraepithelial papillary capillary loop features using narrow band imaging, which is used in diagnosis of epithelial lesions and ranging from benign to malignant. According to the literature sensitivity of NBI in detection malignant lesions (carcinoma in situ or invasive carcinoma) is 88.9%, significantly greater than that of white light visualization (68.9%), specificity of NBI is 93.2% (Ni et al., 2011).

It is possible to expect that using NBI endoscopy will be improved diagnostics early cancerous epithelial changes in hypopharynx and larynx in ENT patients with non-specific symptoms and in cases at the beginning of cancer growth, which is not detected by any other imaging methods. Also using peroperative NBI the investigators expect better detection of resection margin in cancer laser surgery and decrease of re-operations or adjuvant radiotherapy postoperatively.

Aims of project

* to evaluate the value of narrow band imaging in the early detection of laryngeal cancer and its precursor lesions and compare usefulness NBI endoscopy and assessment in standard white light endoscopy
* to carry out detection of epithelial lesions by NBI endoscopy and stroboscopic assessment in patients with changes on the vocal folds and to compare both methods
* to improve detection of precancerous and cancerous changes in hypopharynx and larynx
* to compare extension of mucosal lesions by evaluation of NBI endoscopy and white light endoscopy, and evaluate spreading of cancer in mucosa
* to evaluate influence of extraesophageal reflux (EER) to occurrence of dysplastic lesions

Working hypotheses

1. Precancerous lesions and early mucosal changes are detected in white light endoscopy rarely.
2. Frequency of precancerous lesions and early cancer in hypopharynx and larynx is more often in patients with non-specific symptoms of diseases of head and neck as the investigators thinking.

Methodology

The project is designed as a prospective study which is in compliance with the principles and policies of the Helsinki Declaration and has been approved by the Ethics Committee.

The patients will be enrolled into the study at the phoniatric out-patient part of the ENT department of the University Hospital in Ostrava and ENT department of the University Hospital Hradec Králové. A total of 120-150 patients will be enrolled into the study within 3 years (2012-2015).

Inclusion criteria

1. patients in age 30-80 years
2. patients with chronic inflammation of hypopharynx and larynx longer than 3 months (with pain in throat, globus pharyngeus,…) and/or
3. patients with hoarseness longer than 3 weeks and/or
4. patients with macroscopic laryngeal lesions (leukoplakia, erythroplakia, Reinke oedema, excluded polyps, cystic lesions and nodules)
5. patients with histological confirmation of dysplasia and/or
6. patients with carcinoma in situ/invasive carcinoma of hypopharynx or larynx and/or
7. patients with recurrent respiratory papillomatosis of all ages.

Entry examination Patient enrolled into the study will be asked to complete a questionnaire (age, sex, body weight, smoking habits, alcohol drinking, gastroesophageal/extraesophageal reflux disease in past), to complete Reflux symptom questionnaire (questionnaire used to determine the symptoms typical for EER) and Voice handicap questionnaire. They will undergo endoscopic evaluation of hypopharynx and larynx using flexible white light magnifying videolaryngoscopy with high definition television - lesions will be split according to type of macroscopic pathology (normal mucosa, chronic inflammation, leukoplakia/erythroplakia, papilloma, exophytic tumor, Reinke´s oedema, other), will be evaluated Reflux finding score, videostroboscopy. In narrow band imaging endoscopy will be evaluated epithelial capillary network and classified type of pathological microvasculature. In indicated cases will be performed targeted biopsy in local or general anesthesia.

Data collection, analysis of data and proposal of the statistical processing

The statistical processing will be carried out by Ing. Hana Tomášková, Ph.D. from the Institute of Epidemiology and Public Health, Medical Faculty of the Ostrava University. Suspicion at dysplasia/carcinoma will be compare based on:

1. evaluation of epithelial lesion in white light endoscopy and NBI endoscopy - how many times will be detected malignant lesion in NBI more often than in white light endoscopy
2. evaluation of laryngeal changes in white light endoscopy and videostroboscopy
3. evaluation of laryngeal epithelial changes in NBI endoscopy and videostroboscopy
4. histological evaluation and preoperative endoscopy (white light, NBI, videostroboscopy)
5. connection of EER and benign laryngeal lesion, dysplasia, early stages of carcinoma The methods of descriptive statistics will be used for statistical processing (arithmetic mean, standard deviation, frequency tables), X2 test, Fisher´s exact test, analysis of variance (ANOVA), OR calculation (odds ratio) with 95% confidence intervals and logistic regression. The statistics tests will be assessed on the significance level of 5%. The statistical analysis will be carried out with the Stata v.10 program. The investigators will use the MS Excel program for data collection.

Discussion

Endoscopic evaluation of hypopharyngeal and laryngeal mucosa is new, quite promising method in otorhinolaryngology, which has been established to the praxis 4 years ago. In this method have been examined maximally hundreds of patients. Now is necessary to validate correlation between symptoms of patients and clinical features in different groups of patients, which have non-specific manifestation of upper aero-digestive tract diseases and between patients in different ages. In literature are published reports Japanese gastroenterologists, especially, about impact of NBI endoscopy in diagnosis of epithelial changes. These studies were oriented on esophageal, gastric and intestinal pathologies, but suggest that NBI endoscopy can improve detections of early precancerous and cancerous lesions of hypopharynx and larynx. In case this declaration will be confirmed, in high number of patients with non-specific symptoms could have early diagnosis a strong importance for more successful oncologic treatment.

Benefit of this project in case the investigators confirm the hypothesis that frequency of precancerous lesions and early cancer in hypopharynx and larynx is more often in patients with non-specific symptoms of diseases of head and neck as the investigators thinking and precancerous lesions and early mucosal changes are detected in white light endoscopy rarely, it is possible to expect that the NBI method will be used more often for detection of early cancer in upper aero-digestive tract. This will improve the effect of oncologic treatment and quality of life of these patients.

Intervention

Standard white light magnifying endoscopy, Narrow Band Imaging endoscopy, videostroboscopy, pH monitoring

- see details in "detail description of the study" part of the protocol

ELIGIBILITY:
Inclusion Criteria:

* patients in age 30-80 years
* patients with chronic inflammation of hypopharynx and larynx longer than 3 months (with pain in throat, globbus pharyngeal,…) and/or
* patients with hoarseness longer than 3 weeks and/or
* patients with macroscopic laryngeal lesions (leukoplakia, erythroplakia, Reinke oedema, excluded polyps, cystic lesions and nodules)
* patients with histological confirmation of dysplasia and/or
* patients with carcinoma in situ/invasive carcinoma of hypopharynx or larynx and/or
* patients with recurrent respiratory papillomatosis of all ages

Exclusion Criteria:

* inability to undergo endoscopic examination

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-02; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The number of patients with larger extent of the laryngeal lesison on NBI examination when compared to standard white light endoscopy | 3 years
  The extension of mucosal lesions will be assessed by evaluation of NBI endoscopy and white light endoscopy, together with evaluation of spreading of cancer in mucosa. The total number of patients with larger extent of the laryngeal lesion on NBI examination will be determined, in comparison with the results obtained with standard white light endoscopy.
The number of patients with histologically proven laryngeal cancer | 3 years
  Findings on NBI endoscopy will be compared to findings obtained with white light endoscopy; the usefulness of both methods will be assessed. The number of patients with histologically proven laryngeal cancer will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Kominek, MD,PhD,MBA, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

REFERENCES:
- [Background] Watanabe A, Taniguchi M, Tsujie H, Hosokawa M, Fujita M, Sasaki S. The value of narrow band imaging for early detection of laryngeal cancer. Eur Arch Otorhinolaryngol. 2009 Jul;266(7):1017-23. doi: 10.1007/s00405-008-0835-1. Epub 2008 Nov 4. PMID 18982341
- [Background] Ni XG, He S, Xu ZG, Gao L, Lu N, Yuan Z, Lai SQ, Zhang YM, Yi JL, Wang XL, Zhang L, Li XY, Wang GQ. Endoscopic diagnosis of laryngeal cancer and precancerous lesions by narrow band imaging. J Laryngol Otol. 2011 Mar;125(3):288-96. doi: 10.1017/S0022215110002033. Epub 2010 Nov 8. PMID 21054921
- [Background] Piazza C, Dessouky O, Peretti G, Cocco D, De Benedetto L, Nicolai P. Narrow-band imaging: a new tool for evaluation of head and neck squamous cell carcinomas. Review of the literature. Acta Otorhinolaryngol Ital. 2008 Apr;28(2):49-54. PMID 18669067
- [Background] Piazza C, Cocco D, De Benedetto L, Del Bon F, Nicolai P, Peretti G. Narrow band imaging and high definition television in the assessment of laryngeal cancer: a prospective study on 279 patients. Eur Arch Otorhinolaryngol. 2010 Mar;267(3):409-14. doi: 10.1007/s00405-009-1121-6. Epub 2009 Oct 14. PMID 19826829